CLINICAL TRIAL: NCT07178041
Title: Remote Ischaemic Conditioning for Post-surgical Complications in Hip Fracture (RIC-FRACTURE)
Acronym: RIC-FRACTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH23101
Record Dates: First submitted 2025-06-23; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hip Fracture
Keywords: Hip Fracture; Remote ischaemic conditioning
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIC Interventional Arm (Experimental): Participants recruited to this arm will receive a programme of Remote Ischaemic Conditioning for up to 2 weeks following hip fracture, or discharge from hospital or rehabilitation centre.
  Interventions: Procedure: Remote Ischaemic Conditioning

INTERVENTIONS:
Procedure: Remote Ischaemic Conditioning — Brief episodes of reversible ischaemia are applied to a particular tissue or organ by inflating pressure cuffs around arms or legs to above systolic pressures (mmHg). This procedure is performed for periods that avoid physical injury to the limbs, but induce neurohormonal, systemic or vascular changes in the body. In this study, the treatment will be delivered on the upper arm or unaffected leg.

SUMMARY:
Background Hip fracture affects 70,000 people in the United Kingdom (UK) and costs an estimated £1.1 billion per year to the National Health Service (NHS). Key clinical indicators, such as early surgical repair, have been shown to improve patient outcomes, however morbidity and mortality remain extremely high, reflecting the urgent need for novel therapies to enhance outcomes. Common complications include infection, cardiovascular events, falls and venous thromboembolism. Remote Ischaemic Conditioning (RIC) is a treatment whereby a blood pressure cuff is inflated around an arm or leg to above systolic pressures to occlude blood flow to the limb for short periods of time, that do not result in harm, but trigger innate mechanisms that reduce inflammation, improve organ blood flow and improve bone healing. These may be beneficial effects after hip fracture.

Methods This is a single centre, feasibility study; the participants will receive RIC daily for 40 minutes for 10 days during their inpatient stay. Outcome measures relating primarily to safety, tolerability and feasibility will be collected along with compliance with the intervention. Study feasibility will be determined by success criteria based on recruitment, outcome measure assessment compliance with intervention and follow up.

Secondary outcomes including inpatient mortality, inpatient complications, length of inpatient stay, blood pressure, serum inflammatory and stress markers and functional recovery will also be collected at discharge and 3 month follow up.

Results Data collected on safety, tolerability, and feasibility will be presented descriptively and simple analysis of variance will be undertaken on quantitative data such as blood pressure and serum inflammatory and stress markers between baseline and follow up time points. The study will hopefully establish whether this therapy is feasible to deliver after acute hip fracture.

DETAILED DESCRIPTION:
This is a single centre, single arm feasibility study. The team will aim to recruit 12 participants to complete a programme of RIC for up to 2 weeks following hip fracture or until discharge from hospital or rehabilitation centre.

It is not known whether the main potential protective events resulting from RIC occur due to the short-term effects (likely changes in vascular sensitivity, blood flow etc) or the longer-term effects (modulation of inflammation etc that occur through changes in gene expression). However, the team have chosen a dosing strategy that they feel is practical to deliver given the average length of time people spend in hospital after hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged > 18 years)
* Participant has had a hip fracture identified on X-ray or computed tomography (CT) scan.
* Qualifying hip fracture has not occurred more than 7 days prior to enrollment.
* Able to give written informed consent.
* In the opinion of the treating physician would be able to conform to the study protocol and procedures.

Exclusion Criteria:

* History or presence of significant peripheral vascular disease in the limb conditioned.
* History or presence of complex neuropathic pains or peripheral neuropathy in the limb conditioned.
* Presence of lymphoedema in the limb conditioned.
* Presence of skin ulceration to the limb conditioned.
* Uncontrolled arrhythmia, hypertension, diabetes or angina.
* Third degree heart block or progressive heart failure.
* Acute aortic dissection, myocarditis, or pericarditis.
* Acute deep vein thrombosis, pulmonary embolism.
* Suspected or known dissecting aneurysm.
* Stroke or TIA myocardial infarction in the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of RIC in patients who have suffered hip fracture | From enrolment to the end of follow up at 3 months
  This outcome measure will be assessed by review of their clinical data at baseline and daily intervention visits, review of the side effects during the intervention period and reporting of any AE's throughout the study period. Safety will be defined as;
  * No reported SAE's directly related to RIC
  * Unexpected adverse events in less than 1/3 participants
Participant acceptability - Symptom severity scores | From enrolment to end of follow up at 3 months
  This outcome measure will be assessed by review of side effects / adverse events reported to researchers throughout the intervention period. Acceptability will be defined as;
  ● Symptom severity scores of mild or moderate in less than 1/3 of participants able to report symptoms (based on Likert Scale 1-5; 1 representing no issues; 5 representing severe symptoms)
Participant acceptability - Semi-structured interviews | From enrolment to end of follow up at 3 months
  This outcome measure will be reviewed through the qualitative interviews undertaken in a subset of participants. Acceptability will be defined as;
  ● Reports from semi-structured interviews
Compliance to the intervention | From enrolment to end of treatment at 2 weeks
  This outcome measure will be assessed using the patient monitoring diaries. Compliance will be defined as;
  ● More than 80% of intended RIC cycles completed
Study feasibility | From enrolment to end of follow up at 3 months
  This outcome measure will be assessed by review of patient recruitment, completeness of outcome measure assessments recorded and number of follow up assessments completed. Feasibility will be defined as;
  * Four patients recruited within the first 2 months of recruitment
  * >80% of outcome measure assessments recorded and follow up assessments completed.

SECONDARY OUTCOMES:
Clinical Outcomes - Inpatient Mortality | From enrolment to end of follow up at 3 months
  Explore clinical outcomes including Inpatient mortality (n,%)
Clinical Outcomes - Inpatient Length of Stay | From enrolment to end of follow up at 3 months
  Explore clinical outcomes including Inpatient length of stay (days)
Clinical Outcomes - Rate of inpatient complications | From enrolment to end of follow up at 3 months
  Explore clinical outcomes including Rate of inpatient complications: vascular (venous thromboembolism, acute coronary syndromes, stroke, Transient Ischemic Attack (TIA), systemic embolism, heart failure), infections, renal (acute kidney injury - RIFLE), anaemia (Hb drop ≥ 2g/L) (%)
Clinical Outcomes - Blood pressure | From enrolment to end of follow up at 3 months
  Explore clinical outcomes including Blood pressure (mmHg)
Clinical Outcomes - Function at discharge | From enrolment to end of follow up at 3 months
  Explore clinical outcomes including Function at discharge (Barthel Index)
Clinical Outcomes - Discharge destination | From enrolment to end of follow up at 3 months
  Explore clinical outcomes including Discharge destination
Mechanisms of action | From enrolment to end of treatment at 2 weeks
  * Inflammatory marker analysis at baseline and 2 weeks or prior to discharge
  * Serum catecholamines will also be measured at baseline and 2 weeks or prior to discharge as the stress response may play a critical role in inflammatory response to hip fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ali, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom